CLINICAL TRIAL: NCT03222986
Title: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation Institutional Review Board
Brief Title: Sepsis-damaged Organs-double-markers Identification of Organ Failure Using Fluorescent Nanoparticle Tracking Analysis
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 04-XD37-104
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-02

CONDITIONS: Sepsis With Multiple Organ Dysfunction (MOD)
Keywords: sepsis, nanoparticle tracking analysis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis with organ failure: Patients have organ failure
- Sepsis without organ failure: Patients have no organ failure

SUMMARY:
Systematic establishment of exosome proteomics in co-culture medium and clinical sepsis specimens will be done. Ubiquitination-autophagy-apoptosis biomarkers in exosomes will be detected and correlated to specific organ failure in sepsis. The inflammatory process also will be validated by cytokines analysis. NTA double markers identification will be a smart method to understand the exosome subpopulations.

DETAILED DESCRIPTION:
Background: Sepsis, defined as life-threatening organ dysfunction due to a dysregulated host response to infection, continues to be a source of considerable morbidity and mortality. 19 million cases are seen worldwide each year. Many animal sepsis models had found that sepsis induced multiple organ failure. Ubiquitination, autophagy, apoptosis may involve the process of sepsis related multiple organ failure. Mass spectrometry-based proteomics studies in clinical populations and in rodent and mammalian animal models had started with discovered many novel biomarkers of sepsis. Esoxomes had been found in blood or urine presented the signal of autophagy and apoptosis. Recently, nanoparticle tracking analysis (NTA) was used as a new method for direct and real-time analysis of exosomes. These make it possible to study the exosome biomarkers to analyze septic patients with multiple organ failure.

Aims of the study: This research will be the first study not only to set up macrophage co-cultured with human organ cell models for exosomes secretions but also collect purified exosomes in blood and urine from septic patients. Proteomics studies in exosomes from cell culture and clinical specimens. Analyze ubiquitination, autophage, and apoptosis related biomarkers of exosomes by bioinformatics. Use NTA to set up newly diagnostic methods, to judge the specific organ damage of septic patient by exosomes autophagy-apoptosis biomarkers.

Materials and Methods: In 1st year, LPS (lipopolysaccharide) stimulated macrophage co-cultured with human organ cells will be set up. Exosomes will be isolated and purified from different groups. ScFv (single chain fragments of antibody) will be selected for blocking infection related exosome's transmission. The 2nd year, a total of 60 patients with infection and positive culture results will be included, of whom 30 septic patients had at least one organ failure, others will have only infection. All patients included and classified according to the sepsis-3 criteria. Clinical specimens will be collected from August 2017 to July 2019. Exosome will be isolated and purified. Magnetic beads purification, 2D gel electrophoresis, MALDI-TOF, and bioinformatics will be used to analyze proteomics of exosomes and association of organ-specific markers, autophagy, and apoptosis markers. Western blotting will be done to prove the proteins found by proteomics. Cytokines array in blood also confirm and correlate to autophagy. Finally, we will use nanoparticle tracking analysis with double markers identification to understand the exosome subpopulations of specific organ and autophagy-apoptosis biomarkers.

Possible effect: Systematic establishment of exosome proteomics in co-culture medium and clinical sepsis specimens will be done. In vitro study, ScFv exploring will help to block exsomes uptake as a possible therapeutic method. Ubiquitination-autophagy-apoptosis biomarkers in exosomes will be detected and correlated to specific organ failure in sepsis. The inflammatory process also will be validated by cytokines analysis. NTA double markers identification will be a smart method to understand the exosome subpopulations.

ELIGIBILITY:
Inclusion Criteria:

Septic patients will have an "acute change in total SOFA score ≥ 2 points consequent to infection" Sepsis with organ failure Sepsis without organ failure

Exclusion Criteria:

patients who had chronic respiratory failure with ventilator dependence chronic renal failure with regular hemodialysis

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients will be classified according to the sepsis-3 criteria, also treat according to surviving sepsis campaign guidelines. Every enrolled patients will be traced the infection sources with positive culture results. Enrolled septic patients will have an "acute change in total SOFA score ≥ 2 points consequent to infection"
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Ubiquitination-autophagy-apoptosis biomarkers in exosomes will be detected and correlated to specific organ failure in sepsis | within 24 hrs.
  Ubiquitination-autophagy-apoptosis biomarkers in exosomes will be detected and correlated to specific organ failure in sepsis

SECONDARY OUTCOMES:
The inflammatory process also will be validated by cytokines analysis. | within 24 hrs.
  The inflammatory process also will be validated by cytokines analysis.
NTA double markers identification will be a smart method to understand the exosome subpopulations. | within 24 hrs.
  NTA double markers identification will be a smart method to understand the exosome

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Lin Su, PhD, Study Director — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Wen-Lin Su, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Dombrovskiy, V.Y., et al., Rapid increase in hospitalization and mortality rates for severe sepsis in the United States: a trend analysis from 1993 to 2003. Crit Care Med, 2007. 35(5): p. 1244-50. 2. Angus, D.C., et al., Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med, 2001. 29(7): p. 1303-10. 3. Martin, G.S., et al., The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med, 2003. 348(16): p. 1546-54. 4. van Zanten, A.R., The golden hour of antibiotic administration in severe sepsis: avoid a false start striving for gold*. Crit Care Med, 2014. 42(8): p. 1931-2. 5. Duran-Bedolla, J., et al., Sepsis, mitochondrial failure and multiple organ dysfunction. Clin Invest Med, 2014. 37(2): p. E58-69.